CLINICAL TRIAL: NCT06503185
Title: Multimodal PReoperative Exercise to Decrease PostoperAtive Disability, Cancer RecurrencE and Mortality in Older People With Frailty
Brief Title: The PREPARE for Cancer Surgery Study
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20240283-01H
Record Dates: First submitted 2024-05-28; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Surgery-Complications; Cancer; Frailty; Disability Physical
MeSH Terms: conditions — Neoplasms; Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehabilitation: The intervention is a home-based, multimodal exercise prehabilitation program. Exercise was prescribed in one-hour sessions, performed a minimum of three times per week for three weeks, consisting of: 1) strength training, 2) aerobic exercise and 3) flexibility. The intervention group will receive weekly phone calls to gauge adherence, suggest modifications, provide support and track any adverse events.
  Interventions: Behavioral: Prehabilitation
- Control: The control group received the World Health Organization recommendations for physical activity for people greater or equal to the age of 65 years old pamphlet, as well as a guide to healthy eating for older adults.

INTERVENTIONS:
Behavioral: Prehabilitation — The intervention is a home-based, multimodal exercise prehabilitation program. Exercise is prescribed in one-hour sessions, performed a minimum of three times per week for three weeks, consisting of: 1) strength training, 2) aerobic exercise and 3) flexibility. The intervention group will receive weekly phone calls to gauge adherence, suggest modifications, provide support and track any adverse events.
  Groups: Prehabilitation

SUMMARY:
Our team recently closed recruitment for the PREPARE Trial: PReoperative Exercise to decrease PostoperAtive complication Rates and disability scorEs. The trial enrolled a total of 850 participants; 523 of which were recruited locally at The Ottawa Hospital (TOH). Of the 523 enrolled at TOH, 413 patient participants were on the pathway for cancer surgery and have either completed the study or are in follow-up (participants who withdrew from the full study have been excluded from the sample size in this sub-study proposal). Unexpectedly, almost 80% of the PREPARE Trial sample was linked to cancer surgery - most likely because cancer surgeries were prioritized during the pandemic. This provides us with the opportunity, and perhaps the responsibility, to specifically assess oncology related outcomes. We propose to follow this TOH sub-group of oncology patients for five years following their surgical date, by retrospectively collecting clinical and health administrative data at annual timepoints.

DETAILED DESCRIPTION:
Background: Among cancer surgery patients, systematic reviews suggest a 55% relative improvement in cancer free survival after multimodal prehabilitation. Unfortunately, prehabilitation trials have largely excluded individuals living with frailty. Simply put, we urgently require data from multicenter prehabilitation trials testing interventions that: A) support adequate adherence; and B) focus on older people with frailty having cancer surgery.

Research aims:

1. Does participation in home-based, multimodal prehabilitation improve 5-year event free survival among older adults with frailty having cancer surgery?
2. Does participation in home-based, multimodal prehabilitation improve physical recovery as assessed using patient reported disability scores across the first year after surgery among older adults with frailty having cancer surgery?
3. Does participation in home-based, multimodal prehabilitation lead to earlier return to intended oncologic treatment among older adults with frailty having cancer surgery?

Methods:

Design, setting and participants: This is a cancer-specific sub-study of the PREPARE Trial. This will be a retrospective cohort study performed using clinical and health administrative data from the electronic medical record (EPIC). People => 60 years old with frailty (Clinical Frailty Scale score of 4/9) and cancer having major elective non-cardiac surgery (vascular, intrathoracic, intraabdominal, pelvic, ENT) with expected length of stay of => 2 days will be included.

Intervention: Home-based exercise program with demonstrated efficacy, feasibility and acceptability tailored for people with frailty.

Outcomes and sample size: The primary outcome is event free survival (EFS) in the 5 years after surgery. Secondary outcomes include patient-reported disability trajectory in the year after surgery (WHODAS) and return to intended oncologic treatment (RIOT). Tertiary outcomes include measures of function, complications, survival, and resource use.

Based on our sample size and expected event rate, with 413 patients we will have >80% power to detect a HR=0.7 assuming a median time to event of 2.5 years in the control group).

Expertise: Our team features multidisciplinary clinical and methodological experts, nationally representative knowledge users and patient representatives.

Expected Outcomes: This study will allow us to understand whether prehabilitation is an intervention that can improve both oncologic and physical outcomes through improved recovery for this growing demographic of vulnerable older adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥60 years
* Scheduled, or on the pathway, for elective surgery eLOS ≥2 days
* Expected surgery date between 3 and 12 weeks from enrollment
* Clinical Frailty Scale (CFS) score ≥4/9

Exclusion Criteria:

* Inability to speak English or French
* Co-morbidity preventing assessment or understanding of questionnaires
* Unable to be contacted by telephone
* Unwilling to participate in exercise program
* Cardiac, neurological or orthopedic procedure
* Palliative surgery
* Certain cardiovascular conditions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults with frailty having cancer surgery
Sampling Method: Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) in the 5 years after surgery | 5 years
  Event free survival (similar to disease free survival, but more appropriate for scenarios where surgery is planned after randomization, but could be precluded by disease progression) will be defined using US Food and Drug Administration (FDA) criteria as: the time after randomization to the earliest of a) progression of disease that precludes surgery, local or distant recurrence, or death due to any cause.

SECONDARY OUTCOMES:
Patient-reported disability trajectory in the year after surgery measured using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | 1 year after surgery
  WHODAS is a patient-reported disability scale that assesses limitations in six major life domains (i.e., cognition, mobility, self-care, social interaction, life activities, participation in society). Scores will be normalized to a 100-point scale where higher scores indicate higher disability, with a difference of 5-points representing a minimally important difference after surgery.
Return to intended oncologic treatment (RIOT) | at 4 months after surgery
  This outcome is measured as the time from surgery to initiation (or re-initiation) or chemo-, radiation- or immuno-therapy after surgery, and will be retrospectively censored at 4-months after surgery to reflect variable recommended timeframes for initiation of adjuvant therapy across cancer types

OTHER OUTCOMES:
Function- Katz Index of Activities of Daily Living | Day 3, 5, 7 and up to 30 days after surgery
  The Katz Index measures function in activities of daily living (ADL). The ADLs examined are bathing, dressing, toileting, transferring, continence and feeding. If a person is able to perform the ADL independently, they receive 1 point for that activity. If a person is dependent on others to perform the ADL, they receive 0 points for that activity. A score of 6 is high, meaning the person is independent whereas a score of 0 is low, indicating that the person is very dependent.
Function- Falls | Day 3, 5, 7 and up to 30 days after surgery
  Falls will be documented as a way of assessing function.
Function- Health-related quality of life | Day 3, 5, 7 and up to 30 days after surgery
  EQ5D5L will be used to measure health-related quality of life at baseline and in-hospital after surgery. Participants are asked to select one answer under each domain (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Responses range from having no problems with a particular domain to being unable to engage in that particular domain. Participants are asked to identify on a scale of 0-100 how good or bad their health is on that given day (0 being worst health they can imagine, 100 being best health they can imagine).
Complications | Day 3, 5, 7 and up to 30 days after surgery
  Complications will be collected using the Post-Operative Morbidity Survey, a well-validated prospective instrument for identifying in-hospital complications in key organ systems based on objective criteria
Health system- Discharge disposition | 1 year
  Discharge disposition will be prospectively collected. Assess where the participant will be discharged to once out of hospital.
Health system- Readmissions | 1 year
  Readmissions will be prospectively collected. Linkage to administrative data will allow for collection of readmissions in the year after surgery.
Health system- Long-term care admissions | 1 year
  Linkage to administrative data will allow for collection of subsequent long-term care admissions in the year after surgery.
Health system- Emergency department visits | 1 year
  Emergency department visits since hospital discharge will be captured in the year after surgery
Health system- Healthcare system costs | 1 year
  Linkage to administrative data will allow for collection of health system costs in the year after surgery.
Overall survival | 5 years
  Survival will be confirmed through linkage to health administrative data
Participant feedback | Participants are asked to reflect on the program during a call the day before surgery
  A theoretical domains framework participant survey will identify barriers and facilitators to participation in the exercise group. Responses are on a five-point likert scale ranging from "strongly disagree" to "strongly agree", or "never" to "always" depending on the question asked
Safety (Adverse Events) | Pre-surgery
  Falls, cardiac or respiratory events and unplanned healthcare encounters will be collected during the exercise treatment period. Expert adjudication will determine whether they were study-attributable

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I McIsaac, MD,MPH,FRCPC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including data dictionaries, will be available. This includes individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). The Study Protocol, Statistical Analysis Plan and Informed Consent Form will also be made available. Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data. Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to dmcisaac@toh.ca. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to dmcisaac@toh.ca. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.